CLINICAL TRIAL: NCT02794597
Title: Improving Reproductive Health for Women in Opioid Medication-Assisted Treatment (OMAT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-1236; 1R34DA039381-01A1 (NIH)
Record Dates: First submitted 2016-05-31; First posted 2016-06-09 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Contraception
Keywords: Unplanned Pregnancy, long-acting reversible contraception (LARC), medications for opioid use disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opioid Medication-Assisted Treatment only (No Intervention): Usual care - Opioid Medication Assisted Treatment
- Intervention (Experimental): Peer led, behavioral sexual health intervention: Sexual Health Initiative for Navigation and Empowerment (SHINE).
  Interventions: Behavioral: SHINE intervention group

INTERVENTIONS:
Behavioral: SHINE intervention group — Includes all substance treatment services as well as the brief peer-led behavioral intervention focused on contraceptives, reproductive needs, and motivational interviewing: Sexual Health Initiative for Navigation and Empowerment (SHINE).
  Arms: Intervention

SUMMARY:
Recent research suggests that women with substance use disorders may be at a higher risk of unintended pregnancy. There is a paucity of interventions specifically focused on this population. Through using mixed methods, this study proposes to develop a brief peer-led intervention (based on the Health Belief Model) to prevent unintended pregnancies among women entering opioid medication-assisted treatment; to assess acceptability, feasibility and the initial efficacy of the behavioral intervention; and to conduct exploratory analyses to identify the Health Belief Model constructs that are most influential on use of long-acting reversible contraception methods. Future research would include testing the intervention in a larger scale trial and with other populations.

DETAILED DESCRIPTION:
This study aims to develop a reproductive health intervention to prevent unintended pregnancy for women of child-bearing age in opioid medication-assisted treatment (OMAT). It will be conducted in two phases. The first formative phase will employ individual interviews and focus groups with women between the ages of 18 and 44 and in opioid medication-assisted treatment to better understand: pregnancy desires/motivation and perceived susceptibility and severity, contraceptive knowledge, perceived benefits/barriers, self-efficacy, social norms, behaviors, and access to contraception and family planning services, especially related to long-acting reversible contraception. This information, coupled with prior evidence and theory, will be used to develop a brief peer-led behavioral intervention.

In the second phase, we will conduct a randomized controlled trial to assess the acceptability, feasibility and the initial efficacy of the developed intervention. Women will be recruited from two opioid medication-assisted treatment facilities and once they have consented and the baseline survey is completed they will be randomized to either the behavioral intervention or usual care. Participants will complete a baseline, three and six-month post-baseline follow up survey.

For those randomized to the intervention arm, the first session will occur immediately post-consent and baseline, and the second will occur 2-4 weeks post-baseline. A trained peer-educator will deliver the behavioral intervention that will provide accurate, unbiased information about Long Acting Reversible Contraception (intrauterine devices and subdermal implants) and all other contraceptive methods (including effectiveness, advantages, and disadvantages), help women assess their needs (pregnancy desires compared to behavior), and utilize motivational interviewing to empower them to make an informed decision regarding their sexual health. For those that are interested, the peer-educator will connect women to a Denver Health Community Health Clinic or a clinic of their choosing to further explore appropriate birth control methods. The medical clinic will assess the woman and determine and dispense the most appropriate method.

ELIGIBILITY:
Inclusion Criteria:

* Biologically female
* 18-44 years of age
* receiving medications for opioid use disorder at one of two clinic sites
* not currently pregnant or trying to become pregnant and having no known medical reason that could prevent pregnancy
* having sex or intending to have sex with a biological male
* not currently using a LARC method.

Exclusion Criteria:

* Being too intoxicated at the time of the interview or impaired mentally due to physical or psychological problems to the point that they cannot voluntarily consent to participate in the study and/or respond to the interview
* Have a known reason why they will not be available for the intervention or the follow-up interview.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2016-08; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Rinehart, PhD, Principal Investigator — Denver Health and Hospital Authority
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stowell MA, Thomas-Gale T, Jones HE, Binswanger I, Rinehart DJ. Perspectives among women receiving medications for opioid use disorder: Implications for development of a peer navigation intervention to improve access to family planning services. Subst Abus. 2022;43(1):722-732. doi: 10.1080/08897077.2021.2007514. PMID 35100081
- [Derived] Rinehart DJ, Stowell M, Collings A, Durfee MJ, Thomas-Gale T, Jones HE, Binswanger I. Increasing access to family planning services among women receiving medications for opioid use disorder: A pilot randomized trial examining a peer-led navigation intervention. J Subst Abuse Treat. 2021 Jul;126:108318. doi: 10.1016/j.jsat.2021.108318. Epub 2021 Feb 4. PMID 34116817

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care - Opioid Medication Assisted Treatment (OMAT): The current standard of care for patients at these clinics is to conduct point-of-care urine pregnancy testing at treatment intake and refer positives for follow-up and clinical care. At the time of the study, neither program had standard work in place to assess pregnancy desire or contraceptive use, nor to provide information on contraceptive methods or referral to family planning (FP) services.
- Intervention: Peer-led, behavioral sexual health intervention: Sexual Health Initiative for Navigation and Empowerment (SHINE)
  Intervention: a brief peer-led behavioral intervention focused on contraceptives, reproductive needs, and motivational interviewing.
Period: Overall Study
Arm/Group | Usual Care - Opioid Medication Assisted Treatment (OMAT) | Intervention
Started | 63 | 56
Completed | 63 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Care - Opioid Medication Assisted Treatment: The current standard of care for patients at these clinics is to conduct point-of-care urine pregnancy testing at treatment intake and refer positives for follow-up and clinical care. At the time of the study, neither program had standard work in place to assess pregnancy desire or contraceptive use, nor to provide information on contraceptive methods or referral to FP services.
- Intervention: Peer-led, behavioral sexual health intervention
  Intervention: a brief peer-led behavioral intervention focused on contraceptives, reproductive needs, and motivational interviewing.
- Total: Total of all reporting groups
Arm/Group | Usual Care - Opioid Medication Assisted Treatment | Intervention | Total
Number analyzed (Participants) | 63 | 56 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 56 | 119
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (6.5) | 32.0 (6.4) | 32.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 56 | 119
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 15 | 31
  Not Hispanic or Latino | 47 | 41 | 88
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 4 | 5
  White | 57 | 42 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 8 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 56 | 119

OUTCOME MEASURES:

1. Primary Outcome: Family Planning Visit and Long-acting Reversible Contraception Use at Three and Six Month Follow-up by Condition.
Description: Assess initial efficacy (family planning/clinical visits and uptake of birth control, specifically long-acting reversible contraceptives (LARCs) of the SHINE intervention, using baseline/follow up surveys and review of medical records at three and six months. Specifically, the number of participants that were using LARCs and the number of participants who had attended family visits at each time point.
Time Frame: 3 and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care - Opioid Medication Assisted Treatment | Intervention
Number analyzed (Participants) | 63 | 56
Participants
  3 month LARC use (# of participants) | 2 | 7
  6 month LARC use (# of participants; inclusive of entire 6 month period) | 2 | 7
  Family planning visits at 3 months (# of participants who had a visit) | 8 | 17
  Family planning visits at 6 months (# who had a visit; inclusive of entire 6 month period) | 9 | 20

2. Secondary Outcome: Sexual Health Knowledge at Baseline by Intervention Condition.
Description: Assess the impact of the SHINE intervention on overall sexual and reproductive health knowledge at baseline (based on participants who completed the baseline survey). Reported as percentage of questions answered correctly by participants.
Time Frame: Baseline
Population: Participants who completed the baseline survey
Measure: Number; unit: percentage of correct responses
Arm/Group | Usual Care - Opioid Medication Assisted Treatment | Intervention
Number analyzed (Participants) | 63 | 56
percentage of correct responses | 78.4 | 76.2

3. Secondary Outcome: Sexual Health Knowledge at 3 Month Follow-up by Intervention Condition.
Description: Assess the impact of the SHINE intervention on overall sexual and reproductive health knowledge at 3 month follow-up (based on participants who completed the 3 month follow-up survey). Reported as percentage of questions answered correctly by participants.
Time Frame: 3 months
Population: Participants who completed the 3 month follow-up survey
Measure: Number; unit: percentage of correct responses
Arm/Group | Usual Care - Opioid Medication Assisted Treatment | Intervention
Number analyzed (Participants) | 50 | 38
percentage of correct responses | 81.6 | 81.9

4. Secondary Outcome: Sexual Health Knowledge at 6 Month Follow-up by Intervention Condition.
Description: Assess the impact of the SHINE intervention on overall sexual and reproductive health knowledge at 6 month follow-up (based on participants who completed the 6 month follow-up survey). Reported as percentage of questions answered correctly by participants.
Time Frame: 6 months
Population: Participants who completed the 6 month follow-up survey
Measure: Number; unit: percentage of correct responses
Arm/Group | Usual Care - Opioid Medication Assisted Treatment | Intervention
Number analyzed (Participants) | 50 | 39
percentage of correct responses | 81.8 | 83.5

5. Secondary Outcome: Health Belief Model Constructs (Perceived Threat of Pregnancy) at Baseline by Intervention Condition.
Description: Assess the impact of the SHINE intervention on perceived threat of pregnancy at baseline (based on participants who completed the baseline survey). Reported as number of participants who indicated agreement with the statement, "If I do not use birth control and have unprotected sex, I could get pregnant."
Time Frame: Baseline
Population: Participants who completed the baseline survey
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care - Opioid Medication Assisted Treatment | Intervention
Number analyzed (Participants) | 63 | 56
Participants | 59 | 52

6. Secondary Outcome: Health Belief Model Constructs (Perceived Threat of Pregnancy) at 3 Month Follow-up by Intervention Condition.
Description: Assess the impact of the SHINE intervention on perceived threat of pregnancy at 3 month follow-up (based on participants who completed the 3 month follow-up survey). Reported as number of participants who indicated agreement with the statement, "If I do not use birth control and have unprotected sex, I could get pregnant."
Time Frame: 3 months
Population: Participants who completed the 3 month follow-up survey
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care - Opioid Medication Assisted Treatment | Intervention
Number analyzed (Participants) | 50 | 38
Participants | 42 | 34

7. Secondary Outcome: Health Belief Model Constructs (Perceived Threat of Pregnancy) at 6 Month Follow-up by Intervention Condition.
Description: Assess the impact of the SHINE intervention on perceived threat of pregnancy at 6 month follow-up (based on participants who completed the 6 month follow-up survey). Reported as the number of participants who indicated agreement with the statement, "If I do not use birth control and have unprotected sex, I could get pregnant."
Time Frame: 6 months
Population: Participants who completed the 6 month follow-up survey
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care - Opioid Medication Assisted Treatment | Intervention
Number analyzed (Participants) | 50 | 39
Participants | 44 | 37

8. Secondary Outcome: Health Belief Model Constructs (Contraceptive Cost-benefit) at Baseline by Intervention Condition.
Description: Assess the impact of the SHINE intervention on contraceptive cost-benefit at baseline (based on participants who completed the baseline survey). Perceived contraceptive costs and benefits were assessed with 14 items on a five-point scale describing how strongly participants agreed to each statement. The response scale was coded so that a higher score reflected higher benefits and lower costs and was the desired direction over time. Reported as mean overall score (range 0-56).
Time Frame: baseline
Population: Participants who completed the baseline survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care - Opioid Medication Assisted Treatment | Intervention
Number analyzed (Participants) | 63 | 56
score on a scale | 37.6 (8.3) | 35.6 (8.9)

9. Secondary Outcome: Health Belief Model Constructs (Contraceptive Cost-benefit) at 3 Month Follow-up by Intervention Condition.
Description: Assess the impact of the SHINE intervention on contraceptive cost-benefit at 3 month follow-up (based on participants who completed the 3 month follow-up survey). Perceived contraceptive costs and benefits were assessed with 14 items on a five-point scale describing how strongly participants agreed to each statement. The response scale was coded so that a higher score reflected higher benefits and lower costs and was the desired direction over time. Reported as mean overall score (range 0-56).
Time Frame: 3 months
Population: Participants who completed the 3 month follow-up survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care - Opioid Medication Assisted Treatment | Intervention
Number analyzed (Participants) | 50 | 38
score on a scale | 37.9 (7.6) | 40.1 (8.3)

10. Secondary Outcome: Health Belief Model Constructs (Contraceptive Cost-benefit) at 6 Month Follow-up by Intervention Condition.
Description: Assess the impact of the SHINE intervention on contraceptive cost-benefit at 6 month follow-up (based on participants who completed the 6 month follow-up survey). Perceived contraceptive costs and benefits were assessed with 14 items on a five-point scale describing how strongly participants agreed to each statement. The response scale was coded so that a higher score reflected higher benefits and lower costs and was the desired direction over time. Reported as mean overall score (range 0-56).
Time Frame: 6 months
Population: Participants who completed the 6 month follow-up survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care - Opioid Medication Assisted Treatment | Intervention
Number analyzed (Participants) | 50 | 39
score on a scale | 38.7 (8.3) | 41.5 (9.8)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Usual Care - Opioid Medication Assisted Treatment | Intervention
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/56
Other Adverse Events (participants affected / at risk) | 0/63 | 0/56

LIMITATIONS AND CAVEATS:
Larger sample size needed to detect significant differences in long-acting reversible contraceptive use. The primary study site and where we referred participants for family planning services provides access to low-cost sexual health education and contraception, which may not exist elsewhere.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT02794597/Prot_SAP_000.pdf